CLINICAL TRIAL: NCT07373236
Title: Examining the Effect of Endogenous Glucagon-like Peptide-1 on Glucagon Secretion in Type 1 Diabetes
Brief Title: The Effect of Endogenous GLP-1 on Glucagon Secretion in Type 1 Diabetes
Acronym: EX-HYPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asger Lund, MD (Other)
Responsible Party: Sponsor-Investigator, Asger Lund, MD, Associate professor, MD, Ph.D., University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-25032390
Record Dates: First submitted 2025-11-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; GLP-1; Exendin(9-39)NH2; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — exendin (9-39); Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exendin(9-39)NH2 (Active Comparator): GLP-1 antagonist
  Interventions: Drug: exendin(9-39)amide
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: exendin(9-39)amide — GLP-1 antagonist
  Arms: Exendin(9-39)NH2
Drug: Saline (0.9% NaCl) — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Type 1 diabetes is a serious and burdensome disease that carries the risk of severe complications and premature death, partly due to low blood sugar, also called hypoglycaemia. This is a constant threat, as individuals with type 1 diabetes lack the body's natural safeguard against low blood sugar: the hormone glucagon, which is normally released from the pancreas.

Recent research in mice suggests that this missing safeguard may be due to an imbalance in the hormones released from different cells in the pancreas. More specifically, glucagon-like peptide-1 (GLP-1) appears to play a role in the lack of glucagon secretion. By blocking this hormone using the substance exendin(9-39)NH₂, normalization of glucagon release during low blood sugar has been observed in mice with type 1 diabetes.

The present study aims to investigate whether the same mechanism applies in humans with type 1 diabetes. If confirmed, this finding could form the basis for a novel adjunct treatment to insulin therapy and thereby potentially reduce the risk of hypoglycaemia in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Age between 18 and 70 years
* T1D (diagnosed according to the criteria of the World Health Organization) with HbA1c <69 mmol/mol (<8.5%)
* Body mass index between 19 and 30 kg/m2
* T1D duration of 2-30 years
* C-peptide negative (5 gram arginine-stimulated C-peptide ≤100 pmol/l)
* Treatment with a stable basal-bolus or insulin pump regimen for ≥3 months

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Late microvascular complications except mild non-proliferative retinopathy
* Liver disease (Evaluated by alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times normal values) or a history of hepatobiliary disorder
* Kidney disease (serum creatinine above normal range)
* Treatment with any glucose-lowering drugs beside insulin
* Active or recent (within 5 years) malignant disease
* Regular tobacco smoking or use of other nicotine-containing products
* Any condition considered incompatible with participation by the investigators.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological males, only cisgender men.
Enrollment: 12 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
bsAUC Glucagon | 0-135 minutes
  Entire study periode

SECONDARY OUTCOMES:
bsAUC of Glucagon | 30-90 minutes
  Primary endpoint
Total Glucose infused | 90-135 minutes
  Recovery phase glucose infused
Glucose infused (entire period) | 0-135 minutes
  Entire glucose infused
GLP-1 | 0-135 minutes
  Circulating GLP-1
Cortisol | 0-135 minutes
  Cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No